CLINICAL TRIAL: NCT01086046
Title: A Multicentre, Randomized Controlled Study of Blood Clotting After Transcatheter Atrial Septal Defect Closure
Brief Title: Study of Blood Clotting After Transcatheter Atrial Septal Defect Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Collaborators: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jun Qin, A Multicentre, Randomized Controlled Study of Blood Clotting After Transcatheter Atrial Septal Defect Closure, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cstc2009ab5033
Record Dates: First submitted 2010-03-08; First posted 2010-03-12 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Thrombosis
Keywords: platelet; thrombozyme; ASD; Heparin; Enoxaparin
MeSH Terms: conditions — Thrombosis | interventions — Heparin, Low-Molecular-Weight; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin (Active Comparator): Heparin injection 10 IU/kg/hr within 24h
  Interventions: Drug: Low molecular weight heparin
- Low molecular weight heparin (Experimental): Low molecular weight heparin sodium injection 1mg/kg 2 times in 24 hour
  Low molecular weight heparin sodium injection 1mg/kg 2 times per day in 3 days
  Interventions: Drug: Low molecular weight heparin

INTERVENTIONS:
Drug: Low molecular weight heparin — Low molecular weight heparin sodium injection 1mg/kg 2 times in 24 hour
  Low molecular weight heparin sodium injection 1mg/kg 2 times per day in 3 days.
  Other Names: Enoxaparin

SUMMARY:
The purpose of this study is to evaluate blood clots after Percutaneous ASD Closure in different age, sexuality and defective diameter; evaluating the relationship of blood clotting with Occluder, injury of intima and inflammation;comparation of the effect and safety between different anticoagulation after Percutaneous ASD Repair; explore propose an optimal anticoagulation plan.

DETAILED DESCRIPTION:
Atrial septal defect (ASD) is a common clinical congenital heart disease. It is estimated that the congenital heart disease increase in children by about 15 million annual in China , of which ASD accounted for 10% to 15%. Secundum ASD is the most common clinical type of ASD, of which about 70% is suited to tanscatheter close.With the cardiac catheterization advancing and the devices developing in recent years ,the method has gradually replaced open-chest surgical repair to the person with Secundum ASD. At present, the most widely used device is Amplatzer occluder. With the wide ues of the occlur,there has gradually emerged occluder thrombosis after closure.there are much different methods to antiplatelet and anticoagulation，not only in China but also in the world.so we perfom the study to evaluating the blood clotting after Percutaneous ASD Closure in different age, sexuality and defective diameter; evaluating the relationship of blood clotting with Occluder, injury of intima and inflammation;comparation of the effect and safety between different anticoagulation after Percutaneous ASD Repair; explore propose an optimal anticoagulation plan.

ELIGIBILITY:
Inclusion Criteria:

* Age≥3 years
* Diameter of defect≥5mm and increasing volume load of right heart
* ≤36 mm secondary left to right shunt
* The distance between defective edge and coronaria venosus sinus, inferior caval vein, superior vena and pulmonary vein≥ 5 mm, between artrial-ventricular valve≥7 mm
* The diameter of defect>Occluder
* No other cardiac anomalies need surgery intervention

Exclusion Criteria:

* Hypertension
* Coronary artery disease
* Diabetes
* Atrial fibrillation and oral contraceptive medication
* Aspro, clopidogrel and warfarin in 2 weeks.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
A Multicentre, Randomized Controlled Study of Blood Clotting After Percutaneous Atrial Septal Defect closure | within the first 90 days after closure

CONTACTS AND LOCATIONS:
Overall Officials: lan huang, Study Director — Cardiovascular Department, Xinqiao Hospital, the Third Military Medical University
Locations (1):
- Cardiovascular Department, Xinqiao Hospital, the Third Military Medical University, Chongqing, Chongqing Municipality, China